CLINICAL TRIAL: NCT06201455
Title: Efficacy of Phacogoniotomy in Medically-controlled Primary Open-angle Glaucoma With Cataract a Multicenter Non-inferiority Randomized Controlled Trial
Brief Title: Evaluation of Phacogoniotomy in Medically-controlled POAG
Acronym: ECO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: West China Hospital (Other); Chongqing Medical University (Other); The Second Hospital of Anhui Medical University (Other); Handan City Eye Hospital (Unknown); Shijiazhuang People's Hospital (Other); Chengdu First People's Hospital (Other); Guangdong Hospital of Traditional Chinese Medicine, Zhuhai (Unknown); Joint Shantou International Eye Center of Shantou University and the Chinese University of Hong Kong (Other); Huizhou Municipal Central Hospital (Other)
Responsible Party: Principal Investigator, Xiulan Zhang, Principal Investigator, Zhongshan Ophthalmic Center, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023KYPJ268
Record Dates: First submitted 2023-08-27; First posted 2024-01-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Glaucoma, Open-Angle; Cataract Complicated; Goniotomy
Keywords: Glaucoma, Open-Angle; Cataract; Goniotomy; Minimally invasive glaucoma surgery
MeSH Terms: conditions — Glaucoma, Open-Angle; Capsule Opacification; Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEI+GT (Experimental): Experimental group: Phacoemulsification with intraocular lens implantation (PEI) and goniotomy (GT).
  Interventions: Procedure: PEI+GT
- PEI+MED (Active Comparator): Controll group: Phacoemulsification with intraocular lens implantation (PEI) and medication therapy (MED).
  Interventions: Procedure: PEI+MED

INTERVENTIONS:
Procedure: PEI+GT — After a standard phacoemulsification with intraocular lens implantation (PEI) is performed. The viscoelastic substance will be injected into the anterior chamber again to maintain corneal rigidity. The surgical microscope will be adjusted to tilt 35-40° towards the patient's nasal side, and the patient's head position will be adjusted to tilt 35-40° accordingly. A viscoelastic substance will be applied to the corneal surface to facilitate direct visualization of the angle structures under a gonioscope. The Tanito Microhook will be inserted through the main incision into the anterior chamber, and under gonioscopic guidance, the nasal (or inferonasal) trabecular meshwork and the inner wall of Schlemm's canal will be incised, approximately 120° in extent (60° in each direction).
  Arms: PEI+GT
Procedure: PEI+MED — Participants assigned to control group will undergo routine PEI surgery. Postoperatively, the decision to administer anti-glaucoma medication is based on intraocular pressure (IOP) measurements, and the target IOP is set at 16 mmHg. The selection of medications is informed by the Asia Pacific Glaucoma Guidelines (Kugler Publications, 2016), while the target IOP reference is the European Glaucoma Guidelines.
  Arms: PEI+MED

SUMMARY:
The goal of this multicenter non-inferiority randomized controlled trial is to compare the efficacy of phacoemulsification with intraocular lens implantation (PEI) combined with goniotomy (GT) and PEI combined with medical therapy (MED) in the treatment of medically-controlled primary open-angle glaucoma (POAG) with cataract. The main questions it aims to answer are:

* Whether the PEI+GT was non-inferior to PEI+MED with regard to the intraocular pressure lowering effect in medically-controlled POAG.
* Whether the PEI+GT has value of health economics. Participants will be randomized to receive either PEI+GT or PEI+MED, and followed up with a 1-year period as a primary outcome.

DETAILED DESCRIPTION:
Glaucoma is the leading cause of irreversible blindness worldwide, with primary open-angle glaucoma (POAG) remaining the most common subtype.

Although there are various methods to treat POAG, medication remains the first choice. However, medication therapy has several limitations, such as multiple adverse effects, poor compliance, and high costs. Therefore, it is imperative to explore treatment modalities that reduce medication burden and improve patients' quality of life.

Minimally invasive glaucoma surgery (MIGS) has been widely employed in clinical practice in recent years and become the mainstream surgical approach for POAG treatment. Among them, various forms of Schlemm's canal-based procedures, which were commonly known as ab interno trabeculotomy or goniotomy (GT) have garnered clinical significance due to their advantages of simplicity, minimal invasiveness, low complication rates, and rapid recovery. These procedures can also be combined with phacoemulsification with intraocular lens implantation (PEI). Currently, several GT techniques have been reported using different devices with different ranges of incision. The investigators have proved that a 120-degree GT with or with PEI were effective enough to treat patients with POAG with or without cataract, providing a comparable efficacy with 240 or 360 degree GT. The 120-degree is characterized by not only its efficacy, but also its fewer complications, faster procedure and quicker recovery. Although the techniques have been implemented clinically, further research is needed to evaluate their economics value in terms of reducing patient dependence on medication, relieving the economic burden of glaucoma medications, and improving the quality of life.

Therefore, a non-inferiority randomized controlled trial (RCT) will be conducted in medically controlled POAG patients with cataract, comparing PEI+GT to PEI combined with medication therapy (PEI+MED). The trial aims to validate the effectiveness of GT in reducing medication use, lightening the burden on patients, and providing a novel treatment approach.

ELIGIBILITY:
Inclusion Criteria:

1. 40 ≤ Age ≤ 85 years, gender unrestricted.
2. Diagnosed with POAG.
3. Controlled IOP under 1 to 4 topical hypotensive medications, IOP ≤ 24 mmHg
4. Mean deviation (MD) for perimetry ≥ -16dB.
5. Presence of clinically significant cataract and best-corrected visual acuity measured using the ETDRS chart ≤ 0.63.
6. Voluntary participation of the patient in this study, signing an informed consent form, and agreeing to follow-up visits according to the study protocol.

Exclusion Criteria:

1. Any history of intraocular surgery or ocular trauma.
2. Presence of other types of glaucoma, including primary angle-closure glaucoma and various forms of secondary glaucoma (e.g. secondary angle-closure, pigmentary, steroid-induced, angle-recession, neovascular, inflammatory, and pseudoexfoliation syndrome).
3. Presence of severe ocular diseases of various types that affect the acquisition of ocular parameters or interfere with perimetry.
4. Axial length > 28 mm.
5. Monophthalmia (best-corrected visual acuity of the non-study eye < 0.01).
6. Coexistence of severe systemic diseases affecting the entire body.
7. Pregnant or lactating women.

   * If both eyes of a patient meet the criteria, the eye with worse visual acuity will be selected for inclusion.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-09-28 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
IOP at 12 months after surgery. | Postopertive 12 months.
  The intraocular pressure (mmHg) at 12 months after surgery.

SECONDARY OUTCOMES:
Surgery success of surgery | Postoperative 3, 6, 12 months.
  (i) Complete success (%) is defined as the postoperative 5 < IOP ≤ 16 mmHg with no need for IOP-lowering medication, without any vision-threatening complication or need for re-operation.
  (ii) Qualified success (%) is defined as the postoperative 5 < IOP ≤ 16 mmHg regardless of IOP-lowering medication, without any vision-threatening complication or need for re-operation.
Amount of postoperative anti-glaucomatous medications | Postoperative 1, 3, 6, 12 months.
  The amount of postoperative anti-glaucomatous medications will be measured as: types of medication (No.) × time (No.).
Cost-effectiveness associated parameters | Postoperative 12 months.
  Cost-effectiveness associated parameters: cost of surgery and medications; quality-adjusted life year, etc.

OTHER OUTCOMES:
Surgery complications | Postoperative 1, 3, 6, 12 months.
  Incidence of surgery complications.
Visual acuity | Postoperative 1, 3, 6, 12 months.
  Unit: logMAR
Corneal endothelial cell counting | Postoperative 12 months.
  Unit: cells/mm^2
Visual field | Postoperative 12 months.
  Mean deviation (MD) and pattern standard deviation (PSD) using Humphrey perimetery
Optic nerve head morphology and retinal parameters based on optical coherence tomography | Postoperative 12 months.
  Thickness (μm) of peripapillary retinal nerve fiber layer and macular GC-IPL are collected from optical coherence tomography device.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided